CLINICAL TRIAL: NCT04971499
Title: A Study of Dapansutrile Plus Pembrolizumab in Patients With PD-1 Refractory Advanced Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: April Salama, M.D. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor-Investigator, April Salama, M.D., Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108864
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — dapansutrile; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Selection (Experimental): Dapansutrile starting at 500 mg PO BID plus Pembrolizumab 200 mg IV every three weeks. Dose escalation is planned to a maximum of 1000 mg BID of dapansutrile + pembrolizumab.
  Interventions: Drug: Dapansutrile; Drug: Pembrolizumab
- Dose Expansion (Experimental): Dapansutrile at the RP2D plus Pembrolizumab 200 mg IV every three weeks
  Interventions: Drug: Dapansutrile; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Dapansutrile — 500 mg tablet
Drug: Pembrolizumab — Single-use vial containing 100 mg/4 mL of pembrolizumab

SUMMARY:
This phase 1/2 trial will be conducted in two parts. Part 1 (Dose Selection) is designed to find the dose of dapansutrile with acceptable tolerability in combination with pembrolizumab. Part 1 will consist of up to 2 dose selection cohorts to evaluate the safety and tolerability of dapansutrile + pembrolizumab in patients with PD-1 resistant melanoma to find the recommended part 2 dose (RP2D). Part 1 will include a lead-in phase of dapansutrile monotherapy at 500 mg PO BID. At day 15, combination therapy with pembrolizumab will be initiated. Dose escalation is planned to a maximum of 1000 mg BID of dapansutrile + pembrolizumab.

Part 2 (Dose Expansion) is designed to assess preliminary efficacy of dapansutrile + pembrolizumab in PD-1 resistant melanoma. Once all patients in Part 1 have completed 4 weeks of dapansutrile therapy, the expansion phase will start enrolling. Part 2 will also include a 14-day lead-in period of dapansutrile monotherapy at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed melanoma.
2. Has unresectable Stage III or Stage IV melanoma, per AJCC 8th Edition Staging Criteria, not amenable to local therapy.
3. Male or female participants who are at least 18 years of age on the day of signing informed consent
4. Male participants must agree to use a reliable method of contraception (refer to Section 6.4.1) during the treatment period and for at least 120 days after the last dose of study drug and must refrain from donating sperm during this period.
5. Female participants must not be pregnant or breast feeding and meet at least one of the following conditions:

   1. Not a woman of childbearing potential (WOCBP)
   2. A WOCBP must agree to use a reliable method of contraception (refer to Section 6.4.1) during the treatment period and for at least 120 days after the last dose of study treatment.
6. Participants must have received an anti-PD-1/PD-L1 mAb as part of their most recent line of therapy prior to enrollment in the study.
7. Participants must have progressed on or after treatment with an anti-PD-1/PD-L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies in their most recent line of therapy. PD 1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 8 weeks of an anti-PD-1/PD-L1 mAb
   2. Has demonstrated progression after anti-PD-1/PD-L1 mAb therapy as defined by RECIST v.1.1. The initial evidence of progressive disease (PD) is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression (as defined in 7.c)
   3. Progressive disease has been documented within 6 months from the last dose of anti-PD-1/L1 mAb.

   i. Progressive disease must be determined according to iRECIST ii. This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.

   d. Patients who progress while receiving or within 6 months of receiving the last dose of anti-PD-1/L1 mAb in the neoadjuvant or adjuvant setting will be included. Inclusion of patients who progress within 6 months of stopping neoadjuvant or adjuvant anti-PD-1/L1 mAb will be capped at 20% of the total study population. Inclusion of patients who progress while still receiving neoadjuvant or adjuvant anti-PD-1/L1 mAB will not be capped.
8. The participant provides written informed consent for the trial
9. Measurable disease based on RECIST v.1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions

   1. Multiple target lesions will be allowed and will be selected based on standard RECIST criteria.
   2. The following cutaneous lesions will be considered measurable lesions: lesions ≥ 10 mm in longest diameter or multiple melanoma lesions which in aggregate have a longest diameter of ≥ 10 mm, when measured by caliper.
10. Have available archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.

    1. Newly obtained biopsies are preferred to archived tissue, but archived sample can be used at baseline provided that the patient has only had anti-PD-1/L1 based regimen since obtaining the sample.
    2. Biopsies may be taken from any amenable lesion, but it is preferable to use the same lesion throughout.
    3. Biopsy may be taken from previously irradiated lesions only if they have progressed since radiation therapy.
    4. Patient may still be eligible for study if tumor is not amenable to safe biopsy or biopsy is judged by patient or treating physician to not be in their best interest.
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2. Evaluation of ECOG must be performed within 7 days prior to C1D1.
12. Adequate organ function as defined below. Specimens must have been collected within 7 days prior to the start of study treatment:

    1. Absolute neutrophil count (ANC) ≥1500/µL
    2. Platelets ≥100,000/µL
    3. Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
    4. Creatinine OR measured or calculated creatinine clearance (GFR can be used in place of CrCl) ≤1.5 x ULN OR ≥45 mL/min for participant with creatinine levels >1.5 x institutional ULN
    5. Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels > 1.5 x ULN
    6. AST (SGOT) and ALT (SGPT) ≤2.5 x ULN (≤5 x ULN for participants with liver metastases)
    7. International normalized ratio (INR) OR prothrombin time (PT) ≤1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
    8. Activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants NOTE: Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the last 2 weeks NOTE: Creatinine clearance (CrCl) should be calculated per institutional standard
13. Prior adverse events from anticancer therapy must be resolved to ≤ grade 1, with the exception of alopecia or endocrinopathies, which may be on replacement therapy. Prednisone equivalent of ≤ 10 mg is allowed.

Exclusion Criteria:

1. Ocular or mucosal melanoma
2. A WOCBP who is pregnant or breastfeeding or has a positive pregnancy test within 72 hours prior to receiving study treatment
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to starting study treatment
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
5. Has received cytotoxic chemotherapy for melanoma at any point prior to study enrollment
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
7. Has received an additional line of therapy after the PD-1/PD-L1 therapy prior to starting on this study.
8. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug
9. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years

   a. Exception: time requirement does not apply to patients who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers
10. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate, provided the patient is clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
11. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
12. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
13. History of (non-infectious) pneumonitis/ interstitial lung disease that required steroids or has current pneumonitis/ interstitial lung disease
14. Active infection requiring systemic therapy
15. Known history of Human Immunodeficiency Virus (HIV) infection
16. Known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required
17. Has a known history of active TB (Bacillus Tuberculosis)
18. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
19. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
20. Expecting to conceive or father children within the projected duration of study participation, starting with the screening visit through 120 days after the last dose of trial treatment
21. History of allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of AEs (including SAEs and DLTs) as measured by patient interview and medical record review | 90 days after last dose
Objective response rate as measured by the percentage of patients who achieve a partial or complete response per RECIST v1.1 and iRECIST while receiving study therapy. | Up to 2 years

SECONDARY OUTCOMES:
Progression free survival as measured by the number of patients that have not experienced radiographic disease progression | after 6 months
Progression free survival as measured by the number of patients that have not experienced radiographic disease progression | after 12 months
Overall survival as measured by the number of patients who die due to any cause | after 6 months
Overall survival as measured by the number of patients who die due to any cause | after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: April Salama, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with supporting companies and aggregate data will be included in the final publication.
Supporting Information: Study Protocol, SAP, ICF, CSR